CLINICAL TRIAL: NCT04290000
Title: Collection of Biological Samples From Patients Treated With CAR-T Cells for Hematological Malignancies in Montpellier University Hospital
Brief Title: Collection of Biological Samples From Patients Treated With CAR-T Cells for Hematological Malignancies
Acronym: CAR-T BANK
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0345
Record Dates: First submitted 2020-02-17; First posted 2020-02-28 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma and Acute Lymphoblastic Leukemia
Keywords: CAR T-Cell; lymphoma; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (additional tubes) and marrow (quantity taken in addition from the same aspiration) will be collected in addition to those useful for the follow up of the patients at specific points in his treatment and follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- hematological malignancies: hematological malignancies treated with CAR-T Cells
  Interventions: Other: additional biological samples during CAR-T CELL treatment

INTERVENTIONS:
Other: additional biological samples during CAR-T CELL treatment — Blood samples (additional tubes) and marrow (quantity taken in addition from the same aspiration) will be collected in addition to those useful for the follow up of the patients (progress of their disease after treatment with CAR-T Cells) at specific points in his treatment journey.
  The following samples will also be collected during Apheresis and at Car-T Cells reinjection :
  * Apheresis sampling
  * CAR-T Cells collected from bag rinsate
  In case of invasion, a skin biopsy will be made, 2 days and 8 days after the beginning of the CAR T Cell Treatment, during the patient's hospitalization and during a consultation visit in case of therapeutic progression or failure.

SUMMARY:
Development of CAR-T cell against CD19 B lymphoma and Acute Lymphoblastic Leukemia leaded to 2 authorized medication: Yescarta and Kymriah. Despite impressive outcomes in 3 phase II studies, never met in relapsed or refractory diseases, half of the patients don't respond to this treatment.This can be explained by a low expansion, functional alteration or short persistence of infused cells. Determination of reasons for treatment failure is the first step for optimization of this therapeutics. This project aims to bank blood samples from a cohort of patients treated with CAR-T cell for hematological malignancies in Montpellier University Hospital. Clinical data related to samples will be collected. This samples will be used to determine factors influencing efficacy of CAR-T cells treatments.

DETAILED DESCRIPTION:
Development of CAR-T cell against CD19 B lymphoma and Acute Lymphoblastic Leukema leaded to 2 authorized medication: Yescarta and Kymriah. Despite impressive outcomes in 3 phase II studies, never met in relapsed or refractory diseases, half of the patients don't respond to this treatment.This can be explained by a low expansion, functional alteration or short persistance of infused cells. Determination of reasons for treatment failure is the first step for optimization of this therapeutics. This project aims to bank blood samples from a cohort of patients treated with CAR-T cell for hematological malignancies in Montpellier University Hospital. Clinical data related to samples will be collected. This samples will be used to determine factors influencing efficacy of CAR-T cells treatments.

ELIGIBILITY:
Inclusion Criteria:

* patient treated by CAR-T cell at the University Hospital of Montpellier

Exclusion Criteria:

* refusal to sign consent form
* pregnant woman
* major protected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with CAR-T cell for hematological malignancies in Montpellier University Hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2025-09-27 (Estimated); Study Completion 2040-03-27 (Estimated)

PRIMARY OUTCOMES:
Constitution of biological samples from patient treated with CAR T cells | up to 15 years
  The aim is only to collect biological samples. This collection will be used later to determine factors influencing efficacy of CAR-T cells treatments.
  Blood samples (additional tubes) and marrow (quantity taken in addition from the same aspiration) will be collected in addition to those useful for the follow up of the patients at specific points in his treatment and follow up.
  In case of invasion, a skin biopsy will be made, 2 days and 8 days after the beginning of the CAR T Cell Treatment, during the patient's hospitalization and during a consultation visit in case of therapeutic progression or failure.

SECONDARY OUTCOMES:
patient survival | up to 15 years
  assessment of the patient survival

CONTACTS AND LOCATIONS:
Locations (1):
- Département d'hématologie clinique, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided